CLINICAL TRIAL: NCT00705094
Title: Cardiac Function and Cardiovascular Risk Profile in Testicular Cancer Patients
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GU-24167
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Testicular Cancer; Seminoma; Non-seminomatous
Keywords: cardiovascular risk factors; cardiac function; VO2peak; Chemotherapy
MeSH Terms: conditions — Testicular Neoplasms; Seminoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Testicular cancer patients who have received surgery and are scheduled for surveillance
- 2: Testicular cancer patients who have received surgery and are scheduled for chemotherapy

SUMMARY:
For many years, researchers and doctors have studied different kinds of treatments to improve the survival of men with testicular cancer. However, recent research has shown that many years later, men who had testicular cancer appear to be at higher risk for developing heart disease (heart attack or heart failure), especially if they received chemotherapy. Since these studies were done many years after men received treatment, there was no way to know if other factors contributed to the health problems they experienced. This study is being done because it would be helpful to study heart function and cardiovascular disease risk factors of men who have been diagnosed with testicular cancer, before and after they receive chemotherapy treatment compared to men who receive treatment with surgery alone.

DETAILED DESCRIPTION:
The aim of this pilot study is to examine global and regional LV systolic and diastolic function, cardiac output, cardiac reserve, VO2peak and CVD risk profile in males recently diagnosed with testicular cancer treated with surgery alone or surgery and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* surgery and surveillance
* surgery and multi-cycle chemotherapy
* both good and intermediate prognosis seminoma and non-seminomatous germ cell testicular tumors
* Karnofsky performance index > 70%
* no contraindications to cardiopulmonary testing

Exclusion Criteria:

* documented cardiovascular disease or evidence of myocardial ischemia on the incremental exercise (VO2peak) test.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: testicular cancer patients who have recieved surgery and are scheduled for either chemotherapy or surveillance
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haykowsky, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada